CLINICAL TRIAL: NCT01171521
Title: Management of Complex Wounds Using a Constant Tension External Tissue Expander
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment did not meet projections and numerous lost to follow-up
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Brett Crist, Assistant Professor, Co-Director of Trauma Services, Co-Director Trauma Fellowship, Department of Orthopaedic Surgery, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB1162777
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DermaClose Group (Experimental): DermaClose device applied to complex soft-tissue wound, with or without negative pressure wound therapy, and prospectively followed for primary and secondary outcomes for one year.
  Interventions: Device: DermaClose Group

INTERVENTIONS:
Device: DermaClose Group — The DermaClose external tissue expander provides continuous expanding of the skin around a wound until it has stretched enough to suture the wound edges closed.

SUMMARY:
Complex wounds that cannot be closed primarily are at great risk for complications. A new technique utilizing external tissue expansion holds promise in rapidly decreasing wound area. Facilitation of rapid wound closure is critical in preventing wound complications.

Hypothesis:

Using the Dermaclose Wound Management System (Woundcare Technologies, Inc., Chanhassen, MN) in complex wounds not able to be primarily closed will decrease the time to secondary closure and decrease the need for secondary soft tissue coverage procedures, or if secondary soft tissue procedures are required, its use will decrease the size and complexity of the secondary soft tissue procedures.

Null Hypothesis:

The Dermaclose system will not decrease the need, dimensions, or complexity of secondary soft tissue coverage procedures in complex wounds not able to be primarily closed.

DETAILED DESCRIPTION:
Upon IRB approval, 50 patients with complex soft tissue wounds, with or without an associated fracture that cannot be closed primarily will have the Dermaclose device applied and will be prospectively followed for 1 year. The Dermaclose device will be applied according to the manufacturer's guidelines. This device may be combined with the use of Negative Pressure Wound Therapy. Primary and secondary end points that were initially intended to be included are listed below. However, on SF12 and pain outcome measures were collected and reported.

Initially Intended Primary end points (only SF12 collected and reported):

SF12

1. Initial and final wound dimensions
2. Secondary soft tissue coverage procedures
3. Dimensions and type of secondary soft tissue coverage procedures required compared to initial wound dimensions
4. Method of wound closure
5. Days to wound closure
6. Number and types of procedures required for wound closure
7. Infection requiring reoperation
8. Wound dehiscence requiring reoperation

Initially intended Secondary end points (only #3 collected and reported):

1. Superficial wound dehiscence not requiring reoperation
2. Superficial wound infection not requiring reoperation
3. Visual Analog Pain Scale (VAS) with Dermaclose use
4. Use of negative pressure wound therapy
5. Cost-to-benefit ratio of Dermaclose use - hospital days, number of procedures, procedural and hospital costs including device, negative pressure wound therapy costs, and operating room time and associated costs

Patients will be evaluated daily during their inpatient hospital stays for VAS related to the wound for which the Dermaclose device is used. If the Dermaclose device is used on an outpatient basis, the patient will be asked to complete a daily VAS at the same time to monitor pain associated with device use. After hospital discharge, the patients will be evaluated at 2 weeks, 6 weeks, 3 months, 6 months, and 12 months. They will complete an SF-12 as part of the above evaluations. Patients may be evaluated at more frequent intervals if the need arises. Primary and secondary endpoints will be evaluated at each time point.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Has soft tissue wound(s) that are unable to be closed primarily

Exclusion Criteria:

* Age less than 18
* Has wound(s) that can be closed primarily
* Infected wound
* Unable to comply with protocol
* Prior radiation treatment to skin or soft tissues in the area of the wound
* Friable wound margins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-07; Primary Completion 2013-10 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett D. Crist, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Hospital and Clinics, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- DermaClose Group: DermaClose device applied to complex soft-tissue wound, with or without negative pressure wound therapy, and prospectively followed for primary and secondary outcomes for one year.
  DermaClose external tissue expander: The DermaClose external tissue expander provides continuous expanding of the skin around a wound until it has stretched enough to suture the wound edges closed.
Period: Overall Study
Arm/Group | DermaClose Group
Started | 6
Completed | 0
Not Completed | 6
Not completed — Lost to Follow-up | 5
Not completed — screen failure | 1

BASELINE CHARACTERISTICS:
Population: 5 males, 1 female
Arm/Group | DermaClose Group
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life
Description: The SF-12 contains 12 items from the SF-36 Health Survey - . The SF-12 contains one or two items that measure each of the eight concepts included in the SF-36.
  The Quality of Life SF-12 is a scale from 0 - 100, in which 0 = poor functioning and 100 = excellent functioning.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DermaClose Group
Number analyzed (Participants) | 5
units on a scale | 62.2 (2.4)

2. Secondary Outcome: Pain
Description: Visual Analog Pain Scale (VAS) with DermaClose use, and on study wound at 2 weeks, 6 weeks, 3 months, 6 months, and 12 months. The scale goes from 0 to 10 with 0 being no pain and 10 being the most severe pain imaginable. It is a visual analog scale so is continuous data.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DermaClose Group
Number analyzed (Participants) | 5
units on a scale | 3.8 (3.1)

ADVERSE EVENTS:
Arm/Group | DermaClose Group
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
enrollment was less than predicted and no subject completed the intended 12-month followup. Only SF-12 and pain data were collected for enrolled patients. There was also one screen failure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less